CLINICAL TRIAL: NCT02722135
Title: Open-label, Dose-escalating Trial to Evaluate the Tolerability, Toxicity, Safety, Pharmacokinetics, Pharmacodynamics and Activity of Volasertib Added to the Standard Intensive Salvage Chemotherapy Regimen With Liposomal Daunorubicine, Fludarabine and Cytarabine (DNX-FLA) Followed by Fludarabine and Cytarabine (FLA) in Children From 3 Months to Less Than 18 Years of Age With Acute Myeloid Leukaemia After Failure of the Front-line Therapy
Brief Title: A Study to Find a Safe Dose of Volasertib Given in Addition to Standard Salvage Chemotherapy in Children (Age 3 Months to Less Than 18 Years) With Acute Myeloid Leukaemia, in Whom Front-line Chemotherapy Failed
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.28; 2015-004625-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BI 6727

ARMS (1):
- Volasertib (Experimental)
  Interventions: Drug: Volasertib

INTERVENTIONS:
Drug: Volasertib

SUMMARY:
This is an open-label, dose-escalating trial to evaluate the MTD and/or dose to be used for further development by evaluation of DLT in course 1 and the safety of volasertib when added to standard intensive salvage chemotherapy with DNX-FLA in paediatric patients with AML after failure of first-line therapy. Furthermore, data on efficacy and PK/PD of volasertib in paediatric patients with AML when added to standard intensive salvage chemotherapy will be collected.

ELIGIBILITY:
Inclusion criteria:

* Patients 3 months to <18 years of age at the time of informed consent
* Patients with AML after failure of the front-line intensive AML therapy
* Lansky score at screening >=50 for patients from 3 months to <12 years
* Karnofsky score at screening >=50 for patients from 12 to <18 years
* Use of highly effective methods of birth-control, if sexually active
* Parents/legal guardians and patients have given written informed consent and informed assent suitable for the respective age group

Exclusion criteria:

* Down syndrome
* Acute promyelocytic leukaemia and treatment-related AML
* QTc prolongation
* LVSF <30%
* Cardiac disease and/or dysfunction
* Active uncontrolled infection
* HIV infection, acute or chronic hepatitis
* Inadequate lab parameters
* Impaired renal function
* Pregnancy or nursing
* Further exclusion criteria apply

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Determination of the maximal tolerated dose of volasertib or the recommended volasertib dose for further studies in combination with standard salvage therapy in paediatric patients with AML after failure of the front-line intensive chemotherapy regimen | 4 weeks

SECONDARY OUTCOMES:
Anti-leukaemic activity of volasertib in combination with standard salvage therapy | 8 weeks
Event-free survival (EFS) | up to 5 years
Overall survival (OS) | up to 5 years
Number of patients with clinically relevant lab value changes of calcium (hyper- and/or hypocalcaemia) as judged by the investigator and reported as adverse events (Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher) | 8 weeks
Number of patients with changes in cardiac activity (prolonged QTc interval) reported as clinically relevant observations (i.e. Adverse Events) | 8 weeks
Predose concentration of volasertib before administration of second dose | 8 weeks
Area under the concentration-time curve of volasertib | 8 weeks
Terminal half-life of volasertib in plasma | 8 weeks
Maximum concentration of volasertib | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Ghent, Belgium